# BLUEPRINT FOR WELLNESS (BFW) RESEARCH INFORMED CONSENT

TITLE: Wellness Program Outreach and Effectiveness: A Prospective

Evaluation 2024-2026

PROTOCOL NO.: None

WCG IRB Protocol #20243519

SPONSOR: Quest Diagnostics

INVESTIGATOR: Joseph Doyle Jr., PhD

77 Massachusetts Avenue, E62-516 Cambridge, Massachusetts 02139

**United States** 

STUDY-RELATED

PHONE NUMBER(S): 617-452-3761

Your participation in this study is voluntary. You may decide not to participate or you may leave the study at any time. Your decision will not result in any penalty or loss of benefits to which you are otherwise entitled.

If you have questions, concerns, or complaints, or think this research has hurt you, talk to the research team at the phone number(s) listed in this document.

There is a possibility that identifiers might be removed from your private information or biospecimens and then used or distributed for future research studies without your additional informed consent.

Quest Diagnostics and the Quest family of companies are committed to supporting you in making changes and improving your health by offering comprehensive screening tests and employee wellness programs. Research is an important part of how we make new discoveries that guide our employee wellness program options so that we achieve our program goals. Below is a summary of this research study including key information. Please read the entire consent form before deciding if you want to participate.

# Key information:

- The purpose of this research study is to develop new insights into how employee wellness programs, like Blueprint For Wellness (BFW), impacts the health and wellness of our employees and their spouses/domestic partners ("BFW participants").
- You are being invited to join this study because you are a Quest employee or an employee's spouse/domestic partner signing up for BFW.
- If you join this study, you agree to allow Quest Diagnostics to use certain information (like your answers provided to BFW questions, your employment information and your test results) to perform research described in this consent specifically related to employee wellness programs.
- Quest Diagnostics, Pack Health, and the Quest Welfare Plan (medical plan and BFW) will share eligible BFW participants' information with qualified academic researchers from

Massachusetts Institute of Technology (MIT) Sloan School of Management and the Gies College of Business, University of Illinois at Urbana-Champaign or in scientific publications in a way that cannot identify you.

- There is no direct benefit to you for joining this study. Your participation may help advance scientific knowledge about employee wellness programs, which may or may not benefit all Quest BFW participants in the future.
- There are no physical risks to participating, however there is a small risk that someone could learn about your personal information without permission like in the case of a privacy breach.
- Participation in this research is voluntary and you may choose not to participate. Your
  decision not to participate will not be held against you or affect your access to Quest
  Diagnostics products or services, including BFW. You can change your mind about
  participating at any time. If you decide not to participate in this research or withdraw from
  the research, your employment with Quest will not be affected.

You are being asked to participate in research sponsored by your employer, Quest Diagnostics (QUEST). This research is designed to understand the links between participation in employee wellness programs and BFW participant health outcomes. Quest hired academic researchers from the Massachusetts Institute of Technology (MIT) Sloan School of Management and the Gies College of Business, University of Illinois at Urbana-Champaign (RESEARCHERS) to conduct this study. You will not meet or directly talk to the RESEARCHERS during this research study. Instead, the RESEARCHERS will collect and study BFW participant data that does not directly identify individual employees or spouses/domestic partners.

#### How does it work?

If you consent to participate in this research study, you do not need to do anything different from what you normally do to participate in BFW. Information about BFW participants that consent to participate in this research will be shared with the RESEARCHERS. No information that directly identifies you, such as your name or address, would ever be shared with the RESEARCHERS. The RESEARCHERS will analyze data they receive about:

- How BFW program service providers offer services to BFW participants,
- Limited employment data about employees that cannot individually identify a specific employee,
- Certain BFW participant health and wellness information (medical and pharmacy claims, BFW lab and health survey data) that cannot individually identify a specific BFW participant, and
- Data Quest uses to make decisions about its employee benefit programs.

#### Where does the data come from?

To understand how employer-sponsored wellness programs impact the health outcomes of BFW participants, the RESEARCHERS will look at BFW information (e.g., your answers provided to BFW questions and lab test results, and health support program enrollment, engagement, and test results) and Welfare Plan information (e.g., medical and pharmacy insurance claims.) Additionally, RESEARCHERS will be provided with certain Quest employment data (e.g., salary class, job classification, leave of absence information, employee location code, start/end dates, etc.). RESEARCHERS will also be provided with your basic demographic information (e.g., age, race, ethnicity, sex).

## How will my privacy be protected?

We will store your data securely. We take a number of steps to protect BFW participants' private data by implementing data protection controls to minimize the risk of inadvertent disclosure of your data. Quest Diagnostics strictly adheres to applicable privacy laws and regulations. All electronic study documents will be stored on password protected computers with limited access, and all paper study documents will be stored in locked cabinets. When RESEARCHERS perform research they will have access to your data, but not to your name or other information that directly identifies you.

Your private information and medical record will be shared with individuals and organizations that conduct or watch over this research, including:

- The research sponsor
- People who work with the research sponsor
- Government agencies
- The Institutional Review Board (IRB) that reviewed this research

Your personal data may be stripped of all direct identifying information and combined with others in in an aggregate format to report on the study findings and conclusions. Aggregate reports allow us to share new insights with other for the purpose of developing and implementing improvements to our employee wellness programs and to establish practice standards for implementing such programs.

## Are there risks involved in the study?

Some of the survey and other questions you are asked may be sensitive and make you uncomfortable. You don't have to answer any questions you don't want to. You may receive information about participation in the wellness program(s) that you don't want to receive. You don't have to continue to receive this information and can opt-out of emails and other forms of communication about the wellness programs, you may ignore these communications, or stop participating in a program at any time.

There is a risk that your data, including your self-reported data and your employment and health information, could become public or seen by someone without permission. This could happen in the case of a data breach. If a data breach happens someone could find out who you are or misuse your information. Quest Diagnostics has policies and procedures in place to minimize the risk of this happening. While we believe the chance of this happening is small, it is not zero.

There may be other risks to participating that we don't know about yet.

#### Benefits:

While there are no direct benefits to you, the findings may enhance future wellness programs. You will not be paid for your participation in this study. Consenting to participate in this study is not related to the money you may save on your 2025 Quest medical plan contributions for participation in BFW. If this research leads to new discoveries or other commercial or data products, you will not receive any profits.

### Alternatives:

Your alternative is not to participate in this study.

Who can I talk to about the study if I still have questions?

For questions about the research, my rights as a participant, or to withdraw from the study, I may contact Nicholas Torsiello at <a href="mailto:BFWResearch@packhealth.com">BFWResearch@packhealth.com</a>.

This research is being overseen by WCG IRB. An IRB is a group of people who perform independent review of research studies. You may talk to them at 855-818-2289 or clientcare@wcgclinical.com if:

- You have questions, concerns, or complaints that are not being answered by the research team.
- You are not getting answers from the research team.
- You cannot reach the research team.
- You want to talk to someone else about the research.
- You have questions about your rights as a research subject.

# Please select one of the options below:

| | I DO want to participate in this study. I consent to participate, and I understand that my |
|---|---|
| participa | tion is voluntary, and I may withdraw at any time without penalty or loss of benefits to |
| which I a | m otherwise entitled. |
| | _I DO NOT want to participate in this study. I do not consent to participate, and I |
| understa | nd that I may still participate in Quest employee wellness programs, such as BFW, withou |
| penalty o | r loss of benefits to which I am otherwise entitled. |

### USE OF LEFTOVER BIOLOGICAL SAMPLES AND RELATED DATA FOR FUTURE RESEARCH

When you provide a biological sample (blood and tissue) for laboratory tests, there is usually leftover biological material that is discarded as medical waste. We are asking you to donate your leftover sample rather than have your leftover sample thrown away. Quest Diagnostics plans to conduct future research that may include assay validations for new tests and collaborations with public health agencies and other researcher to develop new medical products using leftover samples. If you consent, your leftover sample will be stripped of any information that directly identifies you, such as your name or address.

We believe the chance someone will identify you is very small, but the risk may change in the future as people come up with new ways of tracing information. If you consent that your leftover sample can be used, the sample will be stored at a facility called a biobank that specializes in the secure storage of human biological samples. Your samples will be stored for 20 years, or until they are no longer usable. Your samples will never be sold. When the sample can no longer be used the sample will be destroyed.

The samples provided will no longer belong to you. There is no direct benefit to you. Research using your samples may lead to new medical knowledge, tests, treatments, or products that help other in the future. These products could have some financial value. There are no plans to provide financial payment to you should this occur.

Tests done for research purposes are not meant to provide clinical information or help care for you. The results are only important for research. Therefore, the results of tests done with your samples will not be provided to you.

You may withdraw permission to allow indirectly identifiable samples to be used for future research by sending a written request to the program administrator at <u>julia.a.larsen@questdiagnostics.com</u>. Samples that have already been used or shared may not be withdrawn.

Samples that have been stripped of ALL identifiers cannot be destroyed because they can no longer be traced back to you.

You do not have to agree to have your leftover Blueprint for Wellness samples used for future test development and research by Quest Diagnostics. If you decide you do not want to consent to the storage and use of your leftover samples it will not impact your employment or eligibility to enroll into Blueprint for Wellness.

If you have any questions, please contact Julia Larsen at julia.a.larsen@questdiagnostics.com.

Please initial next to "no" or "yes" whether you consent for the following:

| Storage and research: |
|---|
| No, I do not agree to have leftover biological samples stored and used for future research. |